CLINICAL TRIAL: NCT05378217
Title: Clinical Evaluation of the Accuracy of AMR-DetecTool for the Diagnostic of Infections With Multi Drug Resistant (MDR) Bacteria
Brief Title: AMR-DetecTool for the Diagnostic of MDR Bacterial Infections
Acronym: AMR DetecTool
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: EIT Health (Other); NG Biotech (Unknown); Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: APHP200100; 2021-A02176-35 (Other: IDRCB)
Record Dates: First submitted 2022-03-04; First posted 2022-05-18 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-11

CONDITIONS: Bacterial Sensitivity Tests; Antimicrobial Drug Resistance
Keywords: beta-Lactamase Resistance; Carbapenem-Resistant Enterobacteriaceae; Vancomycin Resistance; Immunoassay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AMR LFIA Assay — AMR LFIA will be performed in parallel to routine testing on appropriate sample types retrieved from routine testing : Blood, urine, BronchoAlveolar Lavage (BAL), Tracheal Aspirate (TA), Rectal swab

SUMMARY:
The fight against bacteria is one of the greatest challenges faced by societies, especially with the spread of multi drug resistant (MDR) bacteria. The failure to stop the spread of antimicrobial resistance (AMR) is due to a lack of fast detection methods and proper strategies.

Novel, rapid and reliable detection and characterization tests are an urgent need for differentiating between bacterial and viral infections and identifying AMR, so that the most appropriate treatment can be given in a timely manner.

AMR-DetecTool or NG Detectool is a detection system for the direct detection of AMR in clinical samples. The clinical sample is directly processed and a result indicating if the bacteria are resistant to the most relevant antibiotics is immediately shown.

It allows for a dramatic reduction in the treatment decision time upon sample reception from 24 hours (current workflow) to 15-30 minutes.

DETAILED DESCRIPTION:
The fight against bacteria is one of the greatest challenges faced by societies, especially with the spread of multi drug resistant (MDR) bacteria. Among these, the increasing rate of infections caused by Enterobacteriaceae that produce broad-spectrum β-lactamases (ESBLs) and carbapenemases is a major concern worldwide. Moreover, vancomycin-resistance among Enterococcus faecium isolates is becoming a cause of concern in European countries regardless of the geographical location. This increase is due to several factors:

1. Inappropriate use of antibiotics
2. Too late isolation of the carriers
3. Lack of institutional / hospital level strategies to fight antimicrobial resistance (AMR)
4. High transfer abilities due to plasmid-encoded resistance genes The failure to stop the spread of AMR is due to a lack of fast detection methods and proper strategies. Rapid detection and rapid characterization tests are an urgent need. European One Health Action Plan against AMR (2017) states that novel, rapid and reliable diagnostics are crucial for differentiating between bacterial and viral infections and identifying AMR, so that the most appropriate treatment can be given in a timely manner.

AMR-DetecTool or NG Detectool is a detection system for the direct detection of β-lactamases and carbapenemases in clinical samples. It allows for a dramatic reduction in the treatment decision time upon sample reception from 24 hours (current workflow) to 15-30 minutes. When a clinical sample with infection suspicion is received at the microbiology laboratory, the techniques used to determine which the appropriate antibiotic is needed require the sample to be cultured for 16h-24h. Thanks to the DetecTool the culturing step is avoided as the sample is directly processed and a result indicating if the bacteria are resistant to the most relevant antibiotics is immediately shown.

will be performed in parallel to routine testing on appropriate material of selected samples. No additional samples need to be requested to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years-old
* Informed patient and non-opposition received
* Patients matching with at least one of the following situations:
* With a positive blood culture by Gram-staining. Germ must be identified as a Gram-negative bacteria or a Gram-positive cocci in chain (with a special focus on known Vancomycin-Resistant Enterococci (VRE) carrier)
* With an urinary tract infection >104 leukocytes and positive for bacteria (Gram stain or cytometry)
* High-risk (HR) patient for carbapenemase-producing Enterobacterales (CPE) carriage (repatriated patients, tourist returning from endemic country, patients coming from an endemic hospital (same country), contact patient, former carrier, and local HR patients (Long-Term Care Facility (LTCF), etc…)) who have been sampled a rectal swab for routine testing
* With a bronchoalveolar lavage (BAL) or tracheal aspirate (TA) sample and diagnosed as carrier of any of the targeted resistance genes (10-35% chance to develop a Ventilator-associated pneumonia (VAP) with the MDR bacteria)

Exclusion Criteria:

* Patient participation refusal
* Patient subject to judicial protection measure, under tutorship or curatorship
* Patient not-speaking the language spoken in the country of inclusion and without accompanying translator
* Any different sample from the above 4 mentioned one Pregnant women are not excluded to this non-interventional study, as the study does not result in any change in the standard care received by the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with positive bacterial detection and hospitalized in one of the following wards:
  * Medical ICU
  * Surgical ICU
  * Infectious disease unit
  * Nephrology unit
  * Urology unit
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Estimate the diagnostic accuracy of the NG DetecTool device in two populations: population 1 (CTX-M-multi, Carba 5), population 2 (Van A / B, Acinetobacter baumannii-specific oxacillinases (OXA- Ab)). | AMR Detectool results will be obtained within 30 minutes after the patient is included in the study, and the results will be compared to those of the standard routine techniques, that usually require 48 hours.
  Accuracy indices will be for each whole test and for each enzyme: sensibility, specificity, positive and negative predictive values. The reference will be standard technics used in routine (usual cultures and antibiograms). The list of patients with discrepancies between the two tests will be edited for the laboratory to determine the resistance mechanisms of these strains, using polymerase chain reaction (PCR)and/or whole genome sequencing of the bacteria.

SECONDARY OUTCOMES:
Describe a diagnostic algorithm for the use of AMR-lateral flow immunoassay (LFIA), allowing thus a more efficient cost-saving patient-pathway structure in hospitals. | For the entire study period through study completion, an average of 28 days, without censoring at 28 days if an admission is still ongoing.
  Cost-consequence analyses for the use of AMR LFIA over standard techniques based on time to results, cost, patient management and outcome analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry NAAS, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- Bicêtre hospital, Le Kremlin-Bicêtre, France
- Semmelweis University, Budapest, Hungary
- Hospital Clínic School of Medicine, University of Barcelona, Barcelona, Spain